CLINICAL TRIAL: NCT02090959
Title: A Phase 3 Extension Study of Ataluren (PTC124) in Patients With Nonsense Mutation Dystrophinopathy
Brief Title: An Extension Study of Ataluren (PTC124) in Participants With Nonsense Mutation Dystrophinopathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision due to commercial availability of ataluren.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-020e-DMD
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn
Keywords: Duchenne muscular dystrophy; Dystrophinopathy; Nonsense mutation; Premature stop codon; Becker muscular dystrophy; DMD/BMD; PTC124; Ataluren
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ataluren (Experimental): Participants will receive ataluren suspension orally 3 times a day (TID), 10 milligrams/kilogram (mg/kg) at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for up to 144 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered per the dose and schedule specified in the arm.
  Other Names: PTC124

SUMMARY:
The primary objective of this study is to obtain long term safety data of ataluren in male participants with nonsense mutation dystrophinopathy (who participated and completed a previous Phase 3 study of ataluren [PTC124-GD-020-DMD {NCT01826487}]) to augment the overall safety database. Screening and baseline procedures are structured to avoid a gap in treatment between the double-blind study (PTC124-GD-020-DMD) and this extension study.

This study may be further extended by amendment until either ataluren becomes commercially available or the clinical development of ataluren in duchenne muscular dystrophy (DMD) is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study treatment in the previous Phase 3, double-blind study (PTC124-GD-020-DMD).
* Evidence of signed and dated informed consent/assent document(s) indicating that the participant (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial. Note: If the study candidate is considered a child under local regulation, a parent or legal guardian must provide written consent prior to initiation of study screening procedures and the study candidate may be required to provide written assent. The rules of the responsible Institutional Review Board/Independent Ethic Committee (IRB/IEC) regarding whether 1 or both parents must provide consent and the appropriate ages for obtaining consent and assent from the participant should be followed.
* In participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the period of study drug administration and 6-week follow-up period.
* Willingness and ability to comply with scheduled visits, ataluren administration plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug (Litesse® UltraTM [refined polydextrose], polyethylene glycol 3350, Lutrol® micro F127 [poloxamer 407], mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, Cab-O-Sil® M5P [colloidal silica], and magnesium stearate).
* Ongoing participation in any other therapeutic clinical trial.
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, electrocardiogram (ECG) findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bibbiani, M.D., Study Director — PTC Therapeutics
Locations (58):
- United States (21):
  - University of California, Los Angeles, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Children's Hospital Colorado - Center for Cancer and Blood Disorders, Aurora, Colorado
  - Child Neurology Center of Northwest Florida, Gulf Breeze, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, Division of Endocrinology, Metabolism and Lipid Research, St Louis, Missouri
  - Columbia University College of Physicians & Surgeons, New York, New York
  - Children's Hospital Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Childrens Medical Center Dallas, Texas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital - Childhood Cancer and Blood Disorders, Seattle, Washington
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital, Parkville, Victoria
- UZ Leuven, Leuven, Belgium
- Brazil (2):
  - Universidade Federal do Rio de Janeiro - Instituto de Puericultura e Pediatria Martagao Gesteira, Rio de Janeiro
  - Sao Paulo University -HC/FMUSP, São Paulo
- Aleksandrovska Hospital, Sofia, Bulgaria
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Western Ontario, London, Ontario
- Chile (2):
  - Hospital Luis Calvo Mackenna, Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad Catolica, Santiago
- Czechia (2):
  - University Hospital Brno, Brno
  - Motol University Hospital, Prague
- France (4):
  - Hospital de la Timone, Marseille
  - CHU de Nantes, Nantes
  - Hopital Necker - Enfants Malades, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Universitat Munchen - von Haunersche Kinder Clinic, München
- Hadassah University Hospital, Jerusalem, Israel
- Italy (4):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Bambino Gesu Hospital, Rome
  - U.O. Complessa di Neuropsichiatria Infantile, Rome
  - Policlinico Universitario G. Martino, Sicily
- Medical University of Warsaw, Warsaw, Poland
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitari i Politecnic la Fe, Valencia
- Sweden (2):
  - Queen Silvia Children's Hospital, Gothenburg
  - Astrid Lindgren Childrens Hospital, Stockholm
- CHUV Lausanne, Lausanne, Switzerland
- Turkey (Türkiye) (2):
  - Hacettepe Childrens Hospital, Ankara
  - Erciyes University Faculty of Medicine, Talas/Kayseri
- United Kingdom (3):
  - University College London Institute of Child Health, London
  - Royal Manchester Children's Hospital, Manchester
  - The Newcastle upon Tyne Hospitals, NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thangarajh M, Elfring GL, Trifillis P, McIntosh J, Peltz SW; Ataluren Phase 2b Study Group. The relationship between deficit in digit span and genotype in nonsense mutation Duchenne muscular dystrophy. Neurology. 2018 Sep 25;91(13):e1215-e1219. doi: 10.1212/WNL.0000000000006245. Epub 2018 Aug 22. PMID 30135256
- See also: Related Info — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who successfully completed the double-blind, placebo-controlled Phase 3 study (PTC124-GD-020-DMD [NCT01826487]) were screened for this open-label extension study.
Pre-assignment Details: A total of 221 participants completed the double-blind Phase 3 Study PTC124-GD-020-DMD. Of the 221 participants who completed Study PTC124-GD-020-DMD, 219 participants were enrolled in this open-label extension study and 218 were treated.
Groups:
- Ataluren: Participants received ataluren suspension orally 3 times a day (TID), 10 milligrams/kilogram (mg/kg) at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for up to 144 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 219
As-treated Population (All participants who received at least 1 dose of study drug.) | 218
Completed | 68
Not Completed | 151
Not completed — Withdrawal by Subject | 10
Not completed — Adverse Event | 1
Not completed — Investigator decision | 2
Not completed — Study termination | 6
Not completed — Enrolled but not treated | 1
Not completed — Transfer for compassionate use medicine | 4
Not completed — Move to medical need program | 3
Not completed — Entered in to other study | 34
Not completed — Switched to commercial supply | 88
Not completed — Other than specified | 2

BASELINE CHARACTERISTICS:
Population: As Treated (AT) population included all participants who received at least 1 dose of ataluren treatment in this extension study.
Groups:
- Ataluren: Participants received ataluren suspension orally TID, 10 mg/kg at morning, 10 mg/kg at midday, and 20 mg/kg at evening (total daily dose 40 mg/kg) for up to 144 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 169
  Black | 2
  Asian | 13
  Hispanic | 12
  Other | 8
  Missing | 14
6 Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] — The 6MWD test was performed in a 30 meters long flat corridor, where the participant was instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test. Population: This baseline characteristic was analyzed on ambulatory participants only.
  meters
    number analyzed (Participants) | 198
    (all) | 349.885 (105.7913)
Time to Stand From Supine Position [Mean (Standard Deviation); unit: seconds] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  seconds
    number analyzed (Participants) | 199
    (all) | 13.0 (10.34)
Time to Walk/Run 10 Meters [Mean (Standard Deviation); unit: seconds] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  seconds
    number analyzed (Participants) | 215
    (all) | 9.31 (7.388)
Time to Climb 4 Stairs [Mean (Standard Deviation); unit: seconds] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  seconds
    number analyzed (Participants) | 203
    (all) | 9.03 (8.939)
Time to Descend 4 Stairs [Mean (Standard Deviation); unit: seconds] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  seconds
    number analyzed (Participants) | 204
    (all) | 7.52 (8.401)
North Star Ambulatory Assessment (NSAA) Total Score [Mean (Standard Deviation); unit: units on a scale] — NSAA comprised tests of 17 abilities, such as ability to stand, rise from floor, get from lying to sitting, get from sitting to standing, raise one's head, stand on one's heels, hop, jump, and run. For each activity, a score of 0, 1, or 2 was recorded, with 0 = "unable to achieve independently," 1 = "modified method but achieves goal independent of physical assistance from another," or 2 = "normal- achieves goal without any assistance." Sum of these 17 scores was reported as ordinal total score, which can be transformed to a linear total score from 0 (worst) to 100 (best). Population: This baseline parameter was analyzed on ambulatory participants with a baseline value.
  units on a scale
    number analyzed (Participants) | 195
    (all) | 20.73 (8.513)
Performance Upper Limb (PUL) Total Score [Mean (Standard Deviation); unit: units on a scale] — PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into shoulder (4 items), elbow (9 items), and distal (8 items) level dimensions. Scoring options per item may vary from 0-1 and 0-6, according to performance, with higher values corresponding to better performance. Each dimension was scored separately with a maximum score of 16 for shoulder level, 34 for elbow level, and 24 for distal level. Total score was calculated by adding 3 level scores, with a maximum global score of 74 (total score range = 0-74). Higher score = better outcome. Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  units on a scale
    number analyzed (Participants) | 210
    (all) | 68.7 (4.61)
Percent Predicted Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: percent predicted FVC] — FVC is a standard pulmonary function test. FVC was defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100. Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  percent predicted FVC
    number analyzed (Participants) | 210
    (all) | 59.42 (13.843)
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percent predicted FEV1] — FEV1 is a standard pulmonary function test. FEV1 was defined as the volume of air that can forcibly be blown out in 1 second, after full inspiration in the upright position, measured in liters. Percent predicted FEV1 (in %) = [(observed FEV1)/(predicted FEV1)]*100. Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  percent predicted FEV1
    number analyzed (Participants) | 209
    (all) | 53.76 (12.870)
Peak Expiratory Flow (PEF) [Mean (Standard Deviation); unit: liters/second (L/sec)] — PEF was defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  liters/second (L/sec)
    number analyzed (Participants) | 213
    (all) | 3.36 (1.055)
Peak Cough Flow (PCF) [Mean (Standard Deviation); unit: L/sec] — PCF measures an individual's maximum speed of expiration during cough. Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  L/sec
    number analyzed (Participants) | 194
    (all) | 3.30 (1.139)
Pediatric Outcomes Data Collection Instrument (PODCI) Transfers/Basic Mobility Score [Mean (Standard Deviation); unit: units on a scale] — PODCI includes a Global Functioning Scale and 5 core scales: Upper Extremity & Physical Function,Transfer/Basic Mobility, Sports/Physical Functioning, Pain/Comfort,and Happiness. Following PODCI domains were prespecified in protocol for analysis:Transfers/Basic Mobility domain assesses difficulty experienced in performing routine motor activities in daily life. Each domain was scored from 0 (poor outcome/worse health) to 100 (the highest level of functioning & least pain). Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  units on a scale
    number analyzed (Participants) | 216
    (all) | 74.6 (23.66)
Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  millimeters of mercury (mm Hg)
    Systolic blood pressure: number analyzed (Participants) | 217
    Systolic blood pressure | 106.3 (10.72)
    Diastolic blood pressure: number analyzed (Participants) | 217
    Diastolic blood pressure | 68.6 (11.01)
Pulse Rate [Mean (Standard Deviation); unit: beats/minute] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  beats/minute
    number analyzed (Participants) | 217
    (all) | 97.0 (13.31)
Body Temperature [Mean (Standard Deviation); unit: degrees centigrade] — Population: 'Number analyzed' signifies participants of as-treated population analyzed for this parameter.
  degrees centigrade
    number analyzed (Participants) | 217
    (all) | 36.47 (0.453)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE): any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of AEs: graded per Common Terminology Criteria for AEs (CTCAE), Version 3.0 as Grade 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). Drug-related AEs: AEs with possible, probable, unlikely relationship, or unrelated to study drug. Serious AEs (SAEs): death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention. TEAE: an AE that occurred or worsened in the period extending from first dose of study drug in this study to 6 weeks after last dose of study drug in this study. A summary of other non-serious AEs and all SAEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to 6 weeks post-treatment (Week 150)
Population: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 218
Participants
  Any AEs | 202
  SAEs | 24
  Drug-Related AEs | 44
  AEs Leading to Withdrawal From Study | 1
  Mild AEs | 87
  Moderate AEs | 71
  Severe AEs | 42
  Life-threatening AEs | 2

2. Primary Outcome: Number of Participants With Abnormalities in Clinical Laboratory Parameters
Description: Abnormalities in laboratory variables as pre-defined in protocol for safety-monitoring were: Hepatic (Serum alanine aminotransferase [ALT]: increase of greater than [>] 150 units/liter [U/L] with stable or decrease of creatinine kinese [CK]; Serum glutamyl amino transferase [GGT] [U/L]: Grade 2 [>2.5 - 5.0 * upper limit of normal {ULN}]), renal (Serum cystatin C miiligrams/liter [mg/L] >1.33 - 2.00 mg/L; Serum blood urea nitrogen [UREAN] [millimoles/liter {mmol/L}] greater than or equal to [≥]1.5 - 3.0 * ULN; Urine occult blood: 2+ [Small], 3+ [Moderate], 4+ [Large]), and electrolytes (Serum sodium: low [mmol/L], Grade 3-4 [less than {<}130 mmol/L]; serum potassium: high [mmol/L], Grade 3-4 [>6.0 mmol/L]; and Serum bicarbonate [mmol/L]: Grade 2 [<16 - 11 mmol/L]).
Time Frame: Baseline (Day 1) up to 6 weeks post-treatment (Week 150)
Population: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 218
Participants | 29

3. Secondary Outcome: Change From Baseline in 6MWD at Week 144
Description: The 6MWD test was performed in a 30 meters long flat corridor, where the participant was instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
Time Frame: Baseline, Week 144
Population: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study. Here, 'Overall number of participants analyzed' = participants who had both baseline and post-baseline 6MWD value at specified timepoint.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ataluren
Number analyzed (Participants) | 26
meters | -98.18 (86.604)

4. Secondary Outcome: Change From Baseline in Time to Stand From Supine Position at Week 144
Description: If the time taken to perform this test exceeded 30 seconds or if a participant could not perform this test due to disease progression, a value of 30 seconds was used.
Time Frame: Baseline, Week 144
Population: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study. Here, 'Overall number of participants analyzed' = participants who had both baseline and post-baseline value of this parameter at specified timepoint.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 19
seconds | 5.22 (5.104)

5. Secondary Outcome: Change From Baseline in Time to Walk/Run 10 Meters at Week 144
Description: as for outcome 4
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 27
seconds | 2.29 (1.991)

6. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs at Week 144
Description: as for outcome 4
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 22
seconds | 4.01 (7.260)

7. Secondary Outcome: Change From Baseline in Time to Descend 4 Stairs at Week 144
Description: as for outcome 4
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 22
seconds | 2.45 (5.853)

8. Secondary Outcome: Change From Baseline in Physical Function Total Score as Measured by NSAA at Week 144
Description: Physical function was assessed via the NSAA, a functional scale specifically designed for ambulant Duchenne muscular dystrophy (DMD) participants. The assessment comprised tests for 17 abilities of a participant, such as ability to stand, rise from the floor, get from lying to sitting, get from sitting to standing, raise one's head, stand on one's heels, hop, jump, and run. For each activity, a score of 0, 1, or 2 was recorded, with 0 = "unable to achieve independently," 1 = "modified method but achieves goal independent of physical assistance from another," or 2 = "normal- achieves goal without any assistance." The sum of these scores (except for 'raise one's head' activity score) was reported as the ordinal total score, which was transformed to a linear total score ranging from 0 (worst) to 100 (best). Participants with confirmed loss of ambulation at a particular visit were assigned a score of 0.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 40
units on a scale | -7.95 (5.611)

9. Secondary Outcome: Change From Baseline in PUL Total Score at Week 144
Description: The PUL was used to assess motor performance of the upper limb. The PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into shoulder level (4 items), elbow level (9 items), and distal level (8 items) dimensions. Scoring options per item may not be uniform and may vary from 0-1 and 0-6, according to the performance, with higher values corresponding to better performance. Each dimension was scored separately with a maximum score of 16 for shoulder level, 34 for elbow level, and 24 for distal level. Total score was calculated by adding the 3 level scores, with a maximum global score of 74 (total score range = 0-74). Higher score = better outcome.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 44
units on a scale | -4.0 (7.49)

10. Secondary Outcome: Change From Baseline in Percent Predicted FVC as Measured by Spirometry at Week 144
Description: FVC is a standard pulmonary function test. FVC was defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Percent predicted FVC (in %) = [(observed FVC)/(predicted FVC)]*100.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Ataluren
Number analyzed (Participants) | 63
percent predicted FVC | 3.51 (14.253)

11. Secondary Outcome: Change From Baseline in Percent Predicted FEV1 as Measured by Spirometry at Week 144
Description: FEV1 is a standard pulmonary function test. FEV1 was defined as the volume of air that can forcibly be blown out in 1 second, after full inspiration in the upright position, measured in liters. Percent predicted FEV1 (in %) = [(observed FEV1)/(predicted FEV1)]*100.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Ataluren
Number analyzed (Participants) | 63
percent predicted FEV1 | 1.40 (15.319)

12. Secondary Outcome: Change From Baseline in PEF as Measured by Spirometry at Week 144
Description: PEF was defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Ataluren
Number analyzed (Participants) | 65
L/sec | 0.23 (1.099)

13. Secondary Outcome: Change From Baseline in PCF as Measured by Spirometry at Week 144
Description: PCF measures an individual's maximum speed of expiration during cough.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Ataluren
Number analyzed (Participants) | 57
L/sec | 0.53 (1.281)

14. Secondary Outcome: Change From Baseline in PODCI Transfers/Basic Mobility Score at Week 144
Description: Changes in health-related quality of life (HRQL) were measured via the PODCI questionnaire that has been shown to correlate with disease progression and clinical outcome measures in DMD. PODCI includes a Global Functioning Scale and 5 core scales: Upper Extremity and Physical Function,Transfer/Basic Mobility, Sports/Physical Functioning, Pain/Comfort,and Happiness. The following PODCI domain was prespecified in the protocol for analysis:Transfers/Basic Mobility domain assesses difficulty experienced in performing routine motor activities in daily life. Each domain was scored from 0 to 100, with 0 representing a poor outcome/worse health, while 100 representing the highest level of functioning and least pain.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 65
units on a scale | -29.3 (25.05)

15. Secondary Outcome: Number of Participants With Change From Baseline in Activities of Daily Living and Disease Status at Week 144, as Assessed by a Standardized Survey Administered by Site Personnel
Description: Changes in activities of daily living and disease symptoms were captured via a DMD-specific survey administered by Site personnel. At screening or baseline, the participant and/or parent/caregiver were asked to identify any activities of daily living (for example, ambulation, balance, personal hygiene/grooming, dressing and undressing, self-feeding, using the bathroom, handwriting, school performance, behavior or energy level) or symptoms that were affected by the participant's DMD. At post-baseline visit (Week 144), the same participant and/or parent/caregiver was asked to describe any changes from baseline in those activities of daily living/symptoms, within the following categories: physical functioning; general energy level; cognition/school function; emotional/social functioning; and sleep. Changes from baseline were reported on a 5-point Likert scale: 1 (much better), 2 (slightly better), 3 (unchanged), 4 (slightly worse), or 5 (much worse).
Time Frame: Baseline, Week 144
Population: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study. Here, 'Number analyzed 'signifies participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 218
Participants
  Physical Functioning: Walking: number analyzed (Participants) | 143
  Physical Functioning: Walking: Much better | 6
  Physical Functioning: Walking: Slightly better | 3
  Physical Functioning: Walking: Unchanged | 47
  Physical Functioning: Walking: Slightly worse | 32
  Physical Functioning: Walking: Much worse | 55
  Physical Functioning: Climbing Stairs: number analyzed (Participants) | 141
  Physical Functioning: Climbing Stairs: Much better | 6
  Physical Functioning: Climbing Stairs: Slightly better | 4
  Physical Functioning: Climbing Stairs: Unchanged | 37
  Physical Functioning: Climbing Stairs: Slightly worse | 29
  Physical Functioning: Climbing Stairs: Much worse | 65
  Physical Functioning: Upper Extremity Activity: number analyzed (Participants) | 119
  Physical Functioning: Upper Extremity Activity: Much better | 5
  Physical Functioning: Upper Extremity Activity: Slightly better | 6
  Physical Functioning: Upper Extremity Activity: Unchanged | 75
  Physical Functioning: Upper Extremity Activity: Slightly worse | 21
  Physical Functioning: Upper Extremity Activity: Much worse | 12
  Physical Functioning: Other: number analyzed (Participants) | 62
  Physical Functioning: Other: Much better | 3
  Physical Functioning: Other: Slightly better | 2
  Physical Functioning: Other: Unchanged | 29
  Physical Functioning: Other: Slightly worse | 13
  Physical Functioning: Other: Much worse | 15
  Emotional/Social Functioning: number analyzed (Participants) | 134
  Emotional/Social Functioning: Much better | 13
  Emotional/Social Functioning: Slightly better | 16
  Emotional/Social Functioning: Unchanged | 93
  Emotional/Social Functioning: Slightly worse | 7
  Emotional/Social Functioning: Much worse | 5
  Cognition/Social Functioning: number analyzed (Participants) | 133
  Cognition/Social Functioning: Much better | 9
  Cognition/Social Functioning: Slightly better | 24
  Cognition/Social Functioning: Unchanged | 92
  Cognition/Social Functioning: Slightly worse | 8
  Cognition/Social Functioning: Much worse | 0
  General Energy Level: number analyzed (Participants) | 127
  General Energy Level: Much better | 8
  General Energy Level: Slightly better | 8
  General Energy Level: Unchanged | 82
  General Energy Level: Slightly worse | 21
  General Energy Level: Much worse | 8
  Sleep: number analyzed (Participants) | 128
  Sleep: Much better | 11
  Sleep: Slightly better | 11
  Sleep: Unchanged | 95
  Sleep: Slightly worse | 9
  Sleep: Much worse | 2
  Other: number analyzed (Participants) | 31
  Other: Much better | 2
  Other: Slightly better | 2
  Other: Unchanged | 12
  Other: Slightly worse | 8
  Other: Much worse | 7

16. Secondary Outcome: Ataluren Plasma Concentration
Description: Pre-dose ataluren plasma concentrations prior to morning ataluren administration at each clinic visit was assessed using a validated high performance liquid chromatography with tandem mass spectrometry (HPLC/MS-MS) method.
Time Frame: Pre-dose at Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, and 144
Population: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (μg/mL)
Arm/Group | Ataluren
Number analyzed (Participants) | 218
micrograms/milliliter (μg/mL)
  Week 12: number analyzed (Participants) | 210
  Week 12 | 4.5231 (5.08583)
  Week 24: number analyzed (Participants) | 211
  Week 24 | 4.4817 (5.65883)
  Week 36: number analyzed (Participants) | 205
  Week 36 | 5.1551 (5.67555)
  Week 48: number analyzed (Participants) | 201
  Week 48 | 5.2221 (5.32846)
  Week 60: number analyzed (Participants) | 191
  Week 60 | 5.0396 (5.07812)
  Week 72: number analyzed (Participants) | 180
  Week 72 | 6.0677 (6.05912)
  Week 84: number analyzed (Participants) | 171
  Week 84 | 5.4673 (5.15083)
  Week 96: number analyzed (Participants) | 160
  Week 96 | 5.8870 (5.90954)
  Week 108: number analyzed (Participants) | 133
  Week 108 | 5.5905 (6.48016)
  Week 120: number analyzed (Participants) | 119
  Week 120 | 5.2406 (5.69648)
  Week 132: number analyzed (Participants) | 94
  Week 132 | 6.6729 (7.03882)
  Week 144: number analyzed (Participants) | 66
  Week 144 | 5.3898 (6.28487)

17. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at Week 144
Description: Blood pressure determination was performed with the participant in a sitting position after a 5-minute rest.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ataluren
Number analyzed (Participants) | 68
mmHg
  Systolic blood pressure | 0.8 (11.86)
  Diastolic blood pressure | 1.3 (11.60)

18. Secondary Outcome: Change From Baseline in Pulse Rate at Week 144
Description: Pulse rate determination was performed with the participant in a sitting position after a 5-minute rest.
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Ataluren
Number analyzed (Participants) | 68
beats/minute | -0.9 (13.00)

19. Secondary Outcome: Change From Baseline in Body Temperature at Week 144
Time Frame: Baseline, Week 144
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: degrees centigrade
Arm/Group | Ataluren
Number analyzed (Participants) | 68
degrees centigrade | 0.05 (0.545)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 6 weeks post-treatment (Week 150)
Description: AT population included all participants who received at least 1 dose of ataluren treatment in this extension study.
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 0/218
Serious Adverse Events (participants affected / at risk) | 24/218
Other Adverse Events (participants affected / at risk) | 201/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=218)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 5
Hip fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Adenoiditis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Bradycardia (Cardiac disorders) | 1
Transposition of the great vessels (Congenital, familial and genetic disorders) | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1
Cataract (Eye disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=218)
Ear infection (Infections and infestations) | 11
Gastroenteritis (Infections and infestations) | 18
Influenza (Infections and infestations) | 23
Nasopharyngitis (Infections and infestations) | 57
Upper respiratory tract infection (Infections and infestations) | 28
Fall (Injury, poisoning and procedural complications) | 48
Ligament sprain (Injury, poisoning and procedural complications) | 19
Disease progression (General disorders) | 56
Pyrexia (General disorders) | 26
Abdominal pain upper (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Headache (Nervous system disorders) | 42
Haematuria (Renal and urinary disorders) | 20

LIMITATIONS AND CAVEATS:
The study was terminated early per Sponsor decision due to commercial availability of ataluren.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT02090959/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT02090959/SAP_001.pdf